CLINICAL TRIAL: NCT00705653
Title: A Phase I Study of CGC-11047 in Subjects With Advanced Refractory Solid Tumors
Brief Title: Study of CGC-11047 (PG-11047) in Subjects With Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47-01-001
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: cancer; advanced cancer; solid tumors; CGC-11047; PG-11047
MeSH Terms: conditions — Neoplasms | interventions — (N(1),N(12))bis(ethyl)-6,7-dehydrospermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PG-11047 (Experimental)
  Interventions: Drug: PG-11047

INTERVENTIONS:
Drug: PG-11047 — PG-11047 will be administered as a 60-minute intravenous infusion on days 1, 8 and 15 of each 28 day cycle. A treatment cycle will be defined as 4 weeks of therapy. The planned minimum treatment schedule is 2 cycles of PG-11047 treatment (8 weeks).

SUMMARY:
This phase I study aims to assess the safety and tolerability of a new drug - PG-11047 - and to establish what happens to the drug once inside the body. An escalating dose of PG-11047 will be investigated in this study and the maximum tolerated dose of the drug will be established.

DETAILED DESCRIPTION:
This is an open-label phase I, dose-escalation safety study in subjects with refractory solid tumors. The primary objectives of the study are to assess the safety, tolerability, and pharmacokinetics of PG-11047. PG-11047 will be administered as a 60-minute intravenous infusion on days 1, 8 and 15 of each 28 day cycle. The planned minimum treatment schedule is 2 cycles (8 weeks) of PG-11047 treatment. Subjects who tolerate treatment may be eligible to receive additional cycles as per investigator's medical judgment. Evaluation of anti-tumor response will be performed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* non-hematological malignancy where standard therapeutic measures do not exist or no longer effective.
* ECOG - 0-2.
* Life expectancy > 3 months.

Exclusion Criteria:

* chemotherapy or radiotherapy within 4 weeks prior to entering the study.
* previous high-dose chemotherapy with autologous allogeneic hematopoietic stem cell transplantation.
* primary brain tumors or active brain metastases
* history of significant or symptomatic cardiac arrhythmia, prior myocardial infarction or evidence of a current significant ventricular conduction abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Cancer Research Centre, Chicago, Illinois, United States

REFERENCES:
- [Derived] Murray Stewart T, Desai AA, Fitzgerald ML, Marton LJ, Casero RA Jr. A phase I dose-escalation study of the polyamine analog PG-11047 in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2020 Jun;85(6):1089-1096. doi: 10.1007/s00280-020-04082-4. Epub 2020 May 23. PMID 32447421
- See also: Progen Pharmaceuticals website — http://www.progen.com.au

RESULTS

PARTICIPANT FLOW:
Groups:
- PG-11047: Multiple-ascending dose of PG-11047 monotherapy. 60 minute infusion on days 1, 8 and 15 of a 28 day cycle. Dosage was escalated from 50 mg to 750 mg
Period: Overall Study
Arm/Group | PG-11047
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PG-11047
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Secondary Outcome: Preliminary Efficacy
Description: As per RECIST Criteria (V 1.0) by radiologic evaluations: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >= 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD), >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: For the purposes of this study, patients were reevaluated radiologically every 8 weeks. In addition to a baseline scan, confirmatory scans were obtained 6-8 weeks following initial documentation of an objective response, when appropriate.
Population: Patients with non-missing overall response
Measure: Number; unit: percentage (of participants)
Arm/Group | PG-11047
Number analyzed (Participants) | 30
percentage (of participants) | 30

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose below one-third of at least 6 subjects (e.g., 2/6, 3/9, 4/12) experienced a Dose-limiting toxicity (DLT).
  Dose-limiting toxicities (DLTs) used to determine the MTD had to occur during cycle 1 of treatment and had to be considered related to PG-11047.
Time Frame: The MTD had to occur during cycle 1 of treatment
Measure: Number; unit: mg
Arm/Group | PG-11047
Number analyzed (Participants) | 46
mg | 610

ADVERSE EVENTS:
Arm/Group | PG-11047
Serious Adverse Events (participants affected / at risk) | 25/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG-11047 (N=46)
Abdominal pain (Gastrointestinal disorders) | 3 (3) — 1 unrelated to PG-11047; 2 unlikely related to PG-11047
Alteration in mental status (Nervous system disorders) | 1 (1) — Unlikely related to PG-11047
Anemia (Blood and lymphatic system disorders) | 2 (2) — 2 possibly related to PG-11047
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) — Probably related to PG-11047
Aspiration pneumonitis (Infections and infestations) | 1 (1) — Unlikely related to PG-11047
Bowel obstruction (Gastrointestinal disorders) | 4 (5) — 1 unrelated to PG-11047; 4 unlikely related to PG-11047
Bradycardia (Cardiac disorders) | 1 (1) — Possibly related to PG-11047
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated to PG-011047
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unlikely related to PG-11047
Confusion (Nervous system disorders) | 1 (1) — Unrelated to PG-11047
Constipation (Gastrointestinal disorders) | 1 (1) — Unrelated to PG-11047
Diarrhea (Gastrointestinal disorders) | 1 (1) — Probably related to PG-11047
Duodenal stricture (Gastrointestinal disorders) | 1 (1) — Unlikely related to PG-11047
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) — 1 unrelated to PG-11047; 4 unlikely related to PG-11047; 2 possibly related to PG-11047
Elevated amylase (Investigations) | 1 (1) — Unrelated to PG-11047
Elevated bilirubin (Investigations) | 1 (2) — 1 unrelated to PG-11047; 1 unlikely related to PG-11047
Elevated lipase (Investigations) | 1 (1) — Unrelated to PG-11047
Fatigue (General disorders) | 1 (1) — Unlikely related to PG-11047
GI bleed (Gastrointestinal disorders) | 1 (1) — Unlikely related to PG-11047
Gram negative bacteremia (Infections and infestations) | 1 (1) — Unlikely related to PG-11047
Infection (Infections and infestations) | 1 (1) — Unlikely related to PG-11047
Nausea (General disorders) | 2 (2) — 2 unlikely related to PG-11047
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to PG-11047
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — 2 unrelated to PG-11047, 1 unlikely related to PG-11047
Pulmonary embolism (Cardiac disorders) | 1 (1) — Unlikely related to PG-11047
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated to PG-11047
Right arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to PG-11047
Vomitting (General disorders) | 2 (3) — 1 unrelated to PG-11047; 2 unlikely related to PG-11047
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG-11047 (N=46)
Constipation (Gastrointestinal disorders) | 3 (3)
Dizziness (General disorders) | 4 (4)
Fatigue (General disorders) | 16 (24)
Hypotension (Cardiac disorders) | 8 (8)
Mucosal Inflammation (Gastrointestinal disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 13 (14)
Paraesthesia Oral (Nervous system disorders) | 3 (3)
Parasethesia (Nervous system disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
anemia (Blood and lymphatic system disorders) | 9 (11)
anorexia (Metabolism and nutrition disorders) | 10 (12)
dysponea (Respiratory, thoracic and mediastinal disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any formal presentation or publication of data collected from this trial will be considered as a joint publication by the investigator(s) and the appropriate personnel of Progen. Authorship will be determined by mutual agreement.